CLINICAL TRIAL: NCT03110055
Title: Pilot Study to Assess the Effect of Grazoprevir/Elbasvir (ZEPATIER™) and Transarterial Chemoembolization (TACE) vs. TACE Alone in Prolonging Survival of Patients With Non-resectable HCV Associated Hepatocellular Carcinoma
Brief Title: the Effect of Grazoprevir/Elbasvir and TACE vs. TACE Alone in Prolonging Survival of Patients With Non-resectable HCV Associated HCC.
Acronym: ZEPATIER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, michal roll, Head of Research and Development department, Principle investigator, MD., Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-16-OS-0702-CTIL
Record Dates: First submitted 2017-02-08; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: HCV, HCC
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination; Medical Records

STUDY DESIGN:
Intervention Model Description: This is a single center, open label, prospective pilot study. The study will enroll 20 HCV genotype 1 cirrhotic patients with advanced and un-resectable HCC who are eligible for TACE. The patients will receive Grazoprevir/Elbasvir anti-viral treatment in accordance with established guidelines together with regular TACE treatments. Follow up will be for up to 24 months from TACE initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV patients with un-resectable HCC (Experimental): HCV genotype 1 (a and b) cirrhotic patients (child pugh A compensated cirrhosis) with advanced and un-resectable HCC who are eligible for TACE . The patients will receive Grazoprevir/Elbasvir and Transarterial Chemoembolization.
  Their outcomes will be compared to the medical records of patients who underwent Transarterial Chemoembolization only, in the past.
  Interventions: Drug: Grazoprevir/Elbasvir; Other: Medical records; Procedure: Transarterial Chemoembolization

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir — anti-viral treatment for HCV
Other: Medical records — Medical records of patients who underwent Transarterial Chemoembolization only, in the past.
Procedure: Transarterial Chemoembolization — A minimally invasive procedure performed in interventional radiology to restrict a tumor's blood supply. Small embolic particles coated with chemotherapeutic drugs are injected selectively through a catheter into an artery directly supplying the tumor. These particles both block the blood supply and induce cytotoxicity, attacking the tumor in several ways.

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer and the second leading cause of cancer-related deaths in the world. Hepatitis C virus (HCV) is the most common underlying cause of cirrhosis and HCC in the western world. Most patients with HCC present with either non-resectable tumor and/or severe underlying liver dysfunction, and are not suitable candidates for curative treatments by resection or transplantation. Thus, for the majority of patients with HCV related HCC, the only option is prolongation of life without a chance for cure. These patients generally have a poor prognosis with a median survival of less than 1 year. Arterial obstruction of branches of the hepatic artery and simultaneous infusion of chemotherapy (Trans-arterial chemo-embolization or TACE) induces ischemic tumor necrosis with a high rate of objective tumor responses (30-60%). Overall, the median survival after TACE for intermediate HCC is about 20 months, an improvement over supportive care. Treatment with Grazoprevir/Elbasvir showed excellent results in phase 3 studies for patients with HCV genotype 1 (a and b) and genotype 4 infection and is approved for HCV treatment in the USA, Europe and Israel. Anti-HCV therapies may influence HCC biology by decreasing inflammation and may thus alter the tumor microenvironment.

DETAILED DESCRIPTION:
Single center, open label, prospective pilot study. The study will include 20 HCV genotype 1 (a and b) cirrhotic patients (Child Pugh A compensated cirrhosis) with advanced, un-resectable HCC who are eligible for TACE. This pilot study will have one arm which will be compared to historical controls. All patients participating in the study will receive Grazoprevir/Elbasvir treatment according to established guidelines together with regular TACE treatments. The historical controls will refer to patients who received regular TACE treatments alone (standard of HCC care). Follow up will be for up to 24 months from TACE initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic HCV genotype 1 (a and b) infection and un-resectable HCC who are eligible for TACE
2. Ages 18-75 years
3. Willing to take part in a clinical trial and have signed an informed consent
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less
5. Child-Pugh liver function class A
6. Patients with expected survival of less than 1 year
7. Adequate hematologic function (plt≥60, 000 /L; Hb≥8.5 g/dl; and INR≤1.7
8. Adequate hepatic function (albumin ≥3.5 g/dl; total bilirubin, ≤2 mg/dl; ALT and AST ≤5 times the upper limit of the normal range)
9. Adequate renal function (serum creatinine ≤1.5 times the upper limit of normal range).

Exclusion Criteria:

1. Patients unwilling to sign the informed consent
2. Patients unwilling or not capable to complete the anti-viral treatment with Grazoprevir/Elbasvir
3. CPT score >7
4. Patients ineligible for TACE
5. Patients with contraindications to elbasvir/grazoprevir
6. Patients suffering from other underlying liver disease (HBV, HIV, PSC, PBC, AIH etc.)
7. Patients with malignancies other than HCC
8. Patients with previous anti-HCC treatment (RFA, TACE, SIRT or sorafenib)
9. Active alcohol or substance use
10. Previous liver transplantations
11. Child Pugh B or C cirrhosis
12. Total serum bilirubin >1.9 mg/dL
13. Extra-hepatic spread (metastases)
14. Pregnant/lactating women, minors and disabled/incapacitated persons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | assessed up to 24 months
  15% or more increase in survival with the combination treatment of Grazoprevir/Elbasvir and TACE vs. historical control of TACE alone; Time Frame: from start of treatment to death from any cause, or last known date of survival
Adverse events and serious adverse events (AEs, SAEs) | 24 months
  will be assessed in all patients receiving at least one dose of a combination therapy, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time to progression (TTP) | Assessed, up to 24 months
  Time from start of treatment until the first documented event of symptomatic progression.
SVR12 rates | 12 weeks after the last actual dose of Grazoprevir/Elbasvir
  : proportion of patients achieving SVR12
Hepatic de-compensation as assessed by clinical end-points | Once a month up to 24 months
  development of ascites, and will undergo repeated liver function tests every 2 weeks to detect CPT increase.

SECONDARY OUTCOMES:
Time to radiologic progression | The time from start of treatment to disease progression, according to mRECIST, assessed up to 24 months.
  a decrease in tumor in 15 % or more of the patients undergoing combination therapy vs. historical control of TACE alone
Disease-control rate | at least 28 days after the first demonstration of that rating on the basis of independent radiologic review
  The percentage of patients who had a best-response rating of complete response, partial response, or stable disease (according to mRECIST) that was maintained for at least 28 days after the first demonstration of that rating on the basis of independent radiologic review
decrease in tumor markers | Screening and 24 months.
  A 50 % decrease in tumor markers in 15 % or more patients undergoing combination therapy vs. TACE alone
quality of life | At screening, and months 3,13,22.
  Assess quality of life as measured by SF-36 questionnaire
Symptom severity score | At screening, and months 3,13,22.
  Assess severity of symptoms as measured by FSHI8 questionnaire